CLINICAL TRIAL: NCT05343065
Title: Safety of a Real-time Continuous Glucose Monitor-based Insulin Bolus Calculator: The "CGM-IBC" Study B
Brief Title: A Continuous Glucose Monitor Based Insulin Bolus Calculator (CGM-IBC) Study B
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Welldoc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: WD002
Record Dates: First submitted 2022-04-16; First posted 2022-04-25 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2022-04

CONDITIONS: Diabetes Mellitus
Keywords: continuous glucose monitor, insulin calculator
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- CGM insulin bolus calculator arm (Experimental): Participants will use the CGM insulin bolus calculator arm
  Interventions: Device: BlueStar 10

INTERVENTIONS:
Device: BlueStar 10 — An app that coaches individuals with diabetes and supports insulin-dosing based on continuous glucose monitor data

SUMMARY:
This study examines the safety of an app-based insulin bolus calculator that utilizes glucose values from a continuous glucose monitor.

DETAILED DESCRIPTION:
Individuals with type 1 diabetes and those with type 2 diabetes who are prescribed bolus insulin must decide on an insulin dose for any given meal. This dose is often based on what they are eating and their glucose value. Insulin bolus calculators may be helpful in recommending an insulin dose. This study examines the safety of an app-based insulin calculator manufactured by Welldoc (Columbia, MD). This app uses the glucose value and trend arrow, in certain circumstances, to recommend a bolus insulin dose. This study is a single arm trial where continuous glucose monitoring metrics such as time in range will be measured before and after the study participants are given the app.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 or type 2 diabetes using the Dexcom G6 continuous glucose monitor

Exclusion Criteria:

* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2022-07-05 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
The percentage of time a participant's glucose value is between 70 and 180 mg/dL will not be inferior to baseline. | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Jean Park, Principal Investigator — Medstar Health Research Institute
Locations (1):
- MedStar Health Research Institute, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No